CLINICAL TRIAL: NCT03970044
Title: Effectiveness of Once-weekly Exenatide (BCise) Plus Dapagliflozin on 24 Hour Glucose Variability Measured by CGM. A Proof of Concept.
Brief Title: Effectiveness of Exenatide Plus Dapagliflozin on 24 Hour Glucose Variability Measured by CGM. A Proof of Concept.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Consano Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCCR-2019-1
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Exenatide 2 mg plus Dapagaliflozin 10 mg (Experimental): Exenatide extended release, 2 mg weekly, injected Dapagliflozin, 10 mg once daily, orally 14 weeks of treatment
  Interventions: Drug: Exenatide 2 MG; Drug: Dapagliflozin 10 MG
- Exenatide 2 mg (Active Comparator): Exenatide extended release, 2 mg weekly, injected 14 weeks of treatment
  Interventions: Drug: Exenatide 2 MG
- Dapagaliflozin 10 mg (Active Comparator): Dapagliflozin, 10 mg once daily, orally 14 weeks of treatment
  Interventions: Drug: Dapagliflozin 10 MG

INTERVENTIONS:
Drug: Exenatide 2 MG — Glucagon-like peptide-1 receptor
  Other Names: Bydureon; Bydureon BCise; Byetta
  Arms: Exenatide 2 mg; Exenatide 2 mg plus Dapagaliflozin 10 mg
Drug: Dapagliflozin 10 MG — sodium-glucose co-transporter 2 (SGLT2) inhibitor
  Other Names: Farxiga 10 MG
  Arms: Dapagaliflozin 10 mg; Exenatide 2 mg plus Dapagaliflozin 10 mg

SUMMARY:
This is a Phase IV, single site, randomized, open-label, parallel study comparing BYDUREON-BCise plus FARXIGA to BYDUREON-BCise alone and FARXIGA alone in patients diagnosed with Type 2 Diabetes Mellitus (T2DM) on a stable dose of metformin alone.

DETAILED DESCRIPTION:
This is a Phase IV, single site, randomized, open-label, 3 treatment group, parallel study comparing BYDUREON-BCiseTM plus FARXIGATM to BYDUREON-BCiseTM alone and FARXIGATM alone in patients diagnosed with Type 2 Diabetes Mellitus (T2DM) on a stable dose of metformin alone.

Patients who meet all inclusion and none of the exclusion criteria will enter a 1-week Lead-in Period, during which patients will be given a blood glucose meter and fitted with a blinded Continuous Glucose Monitor (CGM) and undergo a 14-day CGM assessment.

After the 1-week Lead-in Period, approximately 60 subjects will be randomized at a 1:1:1 ratio to one of three open-label treatment arms to achieve approximately 20 subjects per treatment arm.

The study consists of a 2-week Screening Period, a 1-week Lead-in Period, a 14-week open-label Treatment Period and a 10-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed written consent prior to any tudy specific procedures
* Male or female, age 18 to 75 years
* Diagnosis of T2DM
* HbA1c >7.5% and <12% obtained at Screening
* Treated with a stable dose of metformin alone (>1500 mg/day) or max tolerated dose for at least 8 weeks prior to Screening
* Body mass index (BMI) <45 kg/m2
* Women of childbearing potential (WOCBP), defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy), must agree to use 2 medically accepted, effective methods of birth control (e.g., hormonal contraceptive, barrier contraceptive with additional spermicide, tubal ligation, or an intrauterine device) prior to IP administration and continuing throughout the study and continuing for 10 weeks after the intake of the last dose of IP
* Females who are postmenopausal must have been postmenopausal for >1 year if they wish not to use contraceptives. If postmenopausal status is questionable, the patient's follicle-stimulating hormone level must be checked and must be elevated and consistent with postmenopausal levels (i.e., >40 IU/L); otherwise these patients must agree to use contraceptives listed above
* Males who are sexually active with WOCBP must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 10 weeks following the last intake of IP to prevent pregnancy in a partner

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
* Previous enrolment in the present study
* Participation in a study within 30 days of planned enrolment in this study and at least 5 half-lives of the investigational product (IP) the patient received in a previous study
* Positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of IP
* Women who are pregnant, breastfeeding, or plan to become pregnant during the course of the study
* History of taking OAD medications other than metformin, during the 8 weeks prior to screening, or have been on insulin therapy within 1 year of screening (with the exception of insulin therapy for rescue or use in gestational diabetes)
* Treated with a GLP-1 receptor agonist within 6 months
* Have a condition that is a contraindicated for use of exenatide (Bydureon BCise), dapagliflozin (Farxiga) or metformin per FDA approved prescribing information
* History of diabetic ketoacidosis requiring medical intervention (e.g., emergency room visit and/or hospitalization) within 3 month prior to screening
* An estimated glomerular filtration rate (eGFR <60 mL/min/1.73 m2 at Screening. A one-time repeat measurement is permitted at the discretion of the investigator, if the value is not consistent with prior values
* History of acute pancreatitis associated or not with using an anti-diabetic drug therapy
* Active liver disease and/or significant abnormal liver function defined as AST > 2 x ULN and/or ALT > 2x ULN and /or serum total bilirubin > 2.0 mg/dl
* History of frequent urinary and/or genital mycotic infections as determined by the investigator
* Uncontrolled thyroid disease as determined by the investigator
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Significant cardiovascular history, as determined per Investigator's discretion
* Ingestion of prescription or over-the-counter weight loss medications during the 3 months prior to screening
* Have a known clinically significant gastric emptying abnormality (eg, severe diabetic gastroparesis or gastric outlet obstruction) or have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery (eg, Lap-Band®) or chronically take drugs that directly reduce gastrointestinal motility
* Chronic or repeated intermittent corticosteroid treatment (subjects receiving stable doses of replacement corticosteroid therapy may be enrolled)
* A history of prior amputation, peripheral vascular disease, or diabetic foot ulcers
* History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed
* Any condition or clinically significant abnormality, which in the Investigator's opinion, may render the patient unable to complete the study or which may pose significant risk to the patient or successful completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
MAGE | 14 weeks
  Compare the change in mean amplitude of glucose excursions from baseline to week 14

SECONDARY OUTCOMES:
Fasting Plasma Glucose | 14 weeks
  Change in fasting plasma glucose from baseline to week 14
HbA1c | 14 weeks
  Change in HbA1c from baseline to week 14
Weight | 14 weeks
  Change in weight from baseline to week 14
Blood Pressure | 14 weeks
  Change in blood pressure from baseline to week 14
Blood Glucose Variability | 14 weeks
  Variability in blood glucose from baseline to weeks 4, 10 and 14
24 Hour Mean Blood Glucose | 17 weeks
  Change in 24 mean blood glucose at multiple time points
Blood Glucose Time In Range | 14 weeks
  Measure the proportion of time patients who had plasma glucose measurements of: <70 mg/dL, >70 mg/dL and <180 mg/dL or >180 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Consano Clinical Research, LLC, Shavano Park, Texas, United States

IPD SHARING:
Plan to Share IPD: No